CLINICAL TRIAL: NCT03561649
Title: Prediction of Adalimumab Treatment Response at 6 Months by Combinatorial Analysis of Serum Biomarkers in Biotherapy Naive Spondyloarthritis: Pilot Study
Brief Title: Prediction of Treatment Response at 6 Months by Combinatorial Analysis of Serum Biomarkers in Biotherapy Naive SpA
Acronym: PRESHUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: SINNOVIAL (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 38RC17.378
Record Dates: First submitted 2018-02-15; First posted 2018-06-19 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Spondylitis, Ankylosing
Keywords: TNF inhibitor; Adalimumab; Spondyloarthritis; Biomarkers analysis; Personalized medicine
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adalimumab (Experimental): Adalimumab is not the experimental study drug. This treatment justifies the inclusion of patients and is used in accordance with its marketing authorization.
  The patients will be seen as part of their follow-up consultation in Rheumatology.
  Modality of administration: The baseline visit should take place no more than 4 weeks before the start of adalimumab treatment, 40mg every 2 weeks, subcutaneously, in accordance with Summary of Product Characteristics.
  At baseline and 6 months follow-up visits, a single blood draw for the biomarker dosage will be added to the standard patient health care follow-up. The clinical examination will also be performed at these two visits, and the clinical response will be assessed after 6 months of adalimumab treatment at M6 follow-up visit.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — This trial will be conducted by rheumatologists who can follow patients with SpA and conduct this trial in good conditions and in accordance with regulatory and legal recommendations.

SUMMARY:
The main objective of this trial is to search for biomarkers associated with the success of adalimumab treatment in order to generate an algorithm to predict the response to this treatment at 6 months in spondyloarthritis and to define its metrological properties on this cohort.

The algorithm will allow to better target patients who will have an important benefit/risk ratio for adalimumab treatment.

DETAILED DESCRIPTION:
The general prevalence of spondyloarthritis (SpA) is 0.5% of the Caucasian population and that of ankylosing spondylitis (AS) is 0.3% in France.

First-line treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) is insufficiently effective in more than half of AS patients in hospitals. These patients are then treated with "anti-tumor necrosis factor alpha" (anti-TNFα). The use of these bio-drugs increasing each year, they become a significant public health and economic challenge. Their development is just beginning, because they are among the largest providers of pharmacy innovations.

The two main cost-drivers appear to be, on the most advanced forms of inflammatory rheumatism, the use of appropriate care structures or services and surgery, especially knee and hip surgery. Among patients treated with biotherapy, clinical practice shows that about one-third (33%) will not respond to selected biopharmaceuticals as these biologics are often prescribed empirically, mainly because of the lack of criteria based on scientific evidence and availability of tools able to predict the response or non-response to these molecules.

Until now, there is no algorithm which can predict the response to biotherapies like adalimumab. The aim of this trial is to search for biomarkers associated with the success of adalimumab treatment in order to generate an algorithm predicting the response to this treatment at 6 months for patients with SpA. This algorithm will be set up from patients' biological and clinical data available after 6 months of adalimumab treatment. A number of 50 patients seems to be statistically sufficient to assess the probability of response or non response to adalimumab in SA with the defined algorithm. A logistic regression model will be used by incorporating the set of available variables.

Then it will be necessary to set up a validation study to determine the metrological properties of the algorithm on an independent cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spondyloarthritis validating ASAS or modified New York criteria for which adalimumab treatment is indicated, and performing the pre-biotherapy assessment;
* Between 18 and 70 years old;
* Biotherapy naive;
* Who can be regularly monitored for 6 months;
* Able to take all the treatment;
* Effective contraception for patients of childbearing age (oral contraceptive, intrauterine device, implant, spermicide, surgical sterilization or abstinence) during the study and at least for 5 months after the last injection;
* Able to read and understand the terms of the protocol;
* Having dated and signed the informed consent form of the trial;
* Affiliated to a social security scheme.

Exclusion Criteria:

* Patients having a contraindication to an anti-TNF;
* Surgical operation scheduled during the trial;
* Having difficulty understanding the French language;
* Having impaired upper functions (dementia of Alzheimer type, etc...);
* Psycho-social instability incompatible with regular follow-up (homeless, addictive behavior, history of psychiatric pathology or any other comorbidity which would make a free and informed consent impossible or limit adherence to the protocol);
* Having previously received a biotherapy. There is no other exclusion criteria taking into account prior therapies and the duration of these therapies;
* Described in articles L.1121-5 to L.1121-8 of the Personal Status Code: pregnant, parturient and nursing women; persons in detention by judicial or administrative decision; adults subject to a legal protection order;
* Already participating in interventional research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Measurement of disease activity: AS-DAS (Ankylosing Spondylitis - Disease Activity Score) | 6 months after baseline
  The primary endpoint is the clinically important ASAS response corresponding to a variation in ASDAS CRP ≥ 1.1.

SECONDARY OUTCOMES:
Measurement of BASDAI response (Bath Ankylosing Spondylitis Disease Activity Index) | 6 months after baseline
  The major clinical ASAS response corresponds to a variation in ASDAS CRP (C-reactive protein) ≥ 2,0 and the major clinical BASDAI 50 response.
  The BASDAI 50 response means an improvement of the BASDAI score by 50% or more. C-Reactive Protein (CRP) in mg/l and Erythrocyte Sedimentation Rate (ESR) in mm at the first hour.
Biomarkers analysis for personalized medicine | At baseline and 6 months later
  Blood draw for selected biomarkers analysis (M0): the dosage data will be used to search for biomarkers associated with successful treatment in order to generate an algorithm predicting the response to adalimumab at 6 months, and to define the metrological properties on this cohort.
  Blood draw for selected biomarkers analysis (M6): we know little about the mechanisms underlying the effect of adalimumab treatment at 6 months in spondyloarthritis, particularly on the biomarker profile. In order to identify possible differences in the profile of selected biomarkers between patients treated with adalimumab at 6 months and biotherapy naive patients (at baseline) and to study the individual variations of the response to this treatment, blood samples will also be collected at 6 months. By using proteomic profiles, the analysis and the comparison of predictive factors at M0 and M6 could be very useful.

CONTACTS AND LOCATIONS:
Overall Officials: Athan BAILLET, MD, PHD, Principal Investigator — University Hospital, Grenoble
Locations (5):
- France (5):
  - CH de Belfort, Belfort
  - CHU de Besançon, Besançon
  - CHRU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Échirolles
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaltonen KJ, Virkki LM, Malmivaara A, Konttinen YT, Nordstrom DC, Blom M. Systematic review and meta-analysis of the efficacy and safety of existing TNF blocking agents in treatment of rheumatoid arthritis. PLoS One. 2012;7(1):e30275. doi: 10.1371/journal.pone.0030275. Epub 2012 Jan 17. PMID 22272322
- [Background] Baeten D, Kruithof E, Van den Bosch F, Van den Bossche N, Herssens A, Mielants H, De Keyser F, Veys EM. Systematic safety follow up in a cohort of 107 patients with spondyloarthropathy treated with infliximab: a new perspective on the role of host defence in the pathogenesis of the disease? Ann Rheum Dis. 2003 Sep;62(9):829-34. doi: 10.1136/ard.62.9.829. PMID 12922954
- [Background] Baillet A, Trocme C, Berthier S, Arlotto M, Grange L, Chenau J, Quetant S, Seve M, Berger F, Juvin R, Morel F, Gaudin P. Synovial fluid proteomic fingerprint: S100A8, S100A9 and S100A12 proteins discriminate rheumatoid arthritis from other inflammatory joint diseases. Rheumatology (Oxford). 2010 Apr;49(4):671-82. doi: 10.1093/rheumatology/kep452. Epub 2010 Jan 25. PMID 20100792
- [Background] Brandt J, Khariouzov A, Listing J, Haibel H, Sorensen H, Grassnickel L, Rudwaleit M, Sieper J, Braun J. Six-month results of a double-blind, placebo-controlled trial of etanercept treatment in patients with active ankylosing spondylitis. Arthritis Rheum. 2003 Jun;48(6):1667-75. doi: 10.1002/art.11017. PMID 12794835
- [Background] Braun J, de Keyser F, Brandt J, Mielants H, Sieper J, Veys E. New treatment options in spondyloarthropathies: increasing evidence for significant efficacy of anti-tumor necrosis factor therapy. Curr Opin Rheumatol. 2001 Jul;13(4):245-9. doi: 10.1097/00002281-200107000-00001. PMID 11555723
- [Background] Braun J, Brandt J, Listing J, Zink A, Alten R, Golder W, Gromnica-Ihle E, Kellner H, Krause A, Schneider M, Sorensen H, Zeidler H, Thriene W, Sieper J. Treatment of active ankylosing spondylitis with infliximab: a randomised controlled multicentre trial. Lancet. 2002 Apr 6;359(9313):1187-93. doi: 10.1016/s0140-6736(02)08215-6. PMID 11955536
- [Background] Braun J, Pham T, Sieper J, Davis J, van der Linden S, Dougados M, van der Heijde D; ASAS Working Group. International ASAS consensus statement for the use of anti-tumour necrosis factor agents in patients with ankylosing spondylitis. Ann Rheum Dis. 2003 Sep;62(9):817-24. doi: 10.1136/ard.62.9.817. PMID 12922952
- [Background] Braun J, Sieper J. Biological therapies in the spondyloarthritides--the current state. Rheumatology (Oxford). 2004 Sep;43(9):1072-84. doi: 10.1093/rheumatology/keh205. Epub 2004 Jun 8. PMID 15187239
- [Background] Claudepierre P, Wendling D, Breban M, Goupillle P, Dougados M. Ankylosing spondylitis, spondyloarthropathy, spondyloarthritis, or spondylarthritis: what's in a name? Joint Bone Spine. 2012 Dec;79(6):534-5. doi: 10.1016/j.jbspin.2012.06.003. Epub 2012 Jul 28. No abstract available. PMID 22841580
- [Background] Haibel H, Rudwaleit M, Brandt HC, Grozdanovic Z, Listing J, Kupper H, Braun J, Sieper J. Adalimumab reduces spinal symptoms in active ankylosing spondylitis: clinical and magnetic resonance imaging results of a fifty-two-week open-label trial. Arthritis Rheum. 2006 Feb;54(2):678-81. doi: 10.1002/art.21563. No abstract available. PMID 16447247
- [Background] Hennigan S, Ackermann C, Kavanaugh A. Adalimumab in ankylosing spondylitis: an evidence-based review of its place in therapy. Core Evid. 2008 Jul 31;2(4):295-305. PMID 21221193
- [Background] Kavanaugh A, Klareskog L, van der Heijde D, Li J, Freundlich B, Hooper M. Improvements in clinical response between 12 and 24 weeks in patients with rheumatoid arthritis on etanercept therapy with or without methotrexate. Ann Rheum Dis. 2008 Oct;67(10):1444-7. doi: 10.1136/ard.2008.094524. Epub 2008 Jun 5. PMID 18535115
- [Background] Lyngberg KK, Harreby M, Bentzen H, Frost B, Danneskiold-Samsoe B. Elderly rheumatoid arthritis patients on steroid treatment tolerate physical training without an increase in disease activity. Arch Phys Med Rehabil. 1994 Nov;75(11):1189-95. doi: 10.1016/0003-9993(94)90003-5. PMID 7979927
- [Background] Machado P, Landewe R, Lie E, Kvien TK, Braun J, Baker D, van der Heijde D; Assessment of SpondyloArthritis international Society. Ankylosing Spondylitis Disease Activity Score (ASDAS): defining cut-off values for disease activity states and improvement scores. Ann Rheum Dis. 2011 Jan;70(1):47-53. doi: 10.1136/ard.2010.138594. Epub 2010 Nov 10. PMID 21068095
- [Background] Madland TM, Larsen A, Brun JG. S100 proteins calprotectin and S100A12 are related to radiographic changes rather than disease activity in psoriatic arthritis with low disease activity. J Rheumatol. 2007 Oct;34(10):2089-92. Epub 2007 Sep 1. PMID 17787039
- [Background] McIntosh E. The cost of rheumatoid arthritis. Br J Rheumatol. 1996 Aug;35(8):781-90. doi: 10.1093/rheumatology/35.8.781. PMID 8761194
- [Background] Maksymowych WP. Biomarkers in axial spondyloarthritis. Curr Opin Rheumatol. 2015 Jul;27(4):343-8. doi: 10.1097/BOR.0000000000000180. PMID 26002025
- [Background] Maksymowych WP, Dougados M, van der Heijde D, Sieper J, Braun J, Citera G, Van den Bosch F, Logeart I, Wajdula J, Jones H, Marshall L, Bonin R, Pedersen R, Vlahos B, Kotak S, Bukowski JF. Clinical and MRI responses to etanercept in early non-radiographic axial spondyloarthritis: 48-week results from the EMBARK study. Ann Rheum Dis. 2016 Jul;75(7):1328-35. doi: 10.1136/annrheumdis-2015-207596. Epub 2015 Aug 12. PMID 26269397
- [Background] Mounach A, El Maghraoui A. Efficacy and safety of adalimumab in ankylosing spondylitis. Open Access Rheumatol. 2014 Aug 13;6:83-90. doi: 10.2147/OARRR.S44550. eCollection 2014. PMID 27790037
- [Background] Pham T, van der Heijde D, Calin A, Khan MA, van der Linden S, Bellamy N, Dougados M; ASAS Working Group. Initiation of biological agents in patients with ankylosing spondylitis: results of a Delphi study by the ASAS Group. Ann Rheum Dis. 2003 Sep;62(9):812-6. doi: 10.1136/ard.62.9.812. PMID 12922951
- [Background] Trocme C, Gaudin P, Berthier S, Barro C, Zaoui P, Morel F. Human B lymphocytes synthesize the 92-kDa gelatinase, matrix metalloproteinase-9. J Biol Chem. 1998 Aug 7;273(32):20677-84. doi: 10.1074/jbc.273.32.20677. PMID 9685427
- [Background] Trocme C, Marotte H, Baillet A, Pallot-Prades B, Garin J, Grange L, Miossec P, Tebib J, Berger F, Nissen MJ, Juvin R, Morel F, Gaudin P. Apolipoprotein A-I and platelet factor 4 are biomarkers for infliximab response in rheumatoid arthritis. Ann Rheum Dis. 2009 Aug;68(8):1328-33. doi: 10.1136/ard.2008.093153. Epub 2008 Jul 29. PMID 18664547
- [Background] Van Den Bosch F, Kruithof E, Baeten D, Herssens A, de Keyser F, Mielants H, Veys EM. Randomized double-blind comparison of chimeric monoclonal antibody to tumor necrosis factor alpha (infliximab) versus placebo in active spondylarthropathy. Arthritis Rheum. 2002 Mar;46(3):755-65. doi: 10.1002/art.511. PMID 11920412
- [Background] Wendling D, Claudepierre P, Lohse A, Toussirot E, Breban M. [Therapeutic use of anti-TNF-alpha agents in spondyloarthropathies]. Presse Med. 2003 Oct 4;32(32):1517-24. French. PMID 14534471
- [Background] Yelin E, Wanke LA. An assessment of the annual and long-term direct costs of rheumatoid arthritis: the impact of poor function and functional decline. Arthritis Rheum. 1999 Jun;42(6):1209-18. doi: 10.1002/1529-0131(199906)42:63.0.CO;2-M. PMID 10366114